CLINICAL TRIAL: NCT00000387
Title: Self-Management Therapy for Youth With Schizophrenia
Acronym: FamCent
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Karen G. Schepp, NIMH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH056580 (NIH); DSIR CT-S
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Schizophrenia
Keywords: Adolescence; Family; Female; Human; Male; Schizophrenia; Self Care; Community Health Services
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A,1,III (Experimental): Behavioral intervention - Self management therapy
  Interventions: Behavioral: Self-management therapy
- A,2,III (Active Comparator): Regular treatment
  Interventions: Behavioral: Self-management therapy

INTERVENTIONS:
Behavioral: Self-management therapy — Behavioral
Behavioral: Self-management therapy

SUMMARY:
The purpose of this study is to test the effectiveness of a family-centered, community-based, self-management intervention (Self-Management Therapy) for adolescents with schizophrenia. The study will test the intervention's effectiveness in improving the adolescents' behavior, thinking, mood, and use of substances such as drugs and alcohol. The study also will look at the effects of the patient on the family.

The intervention involves training in recognizing symptoms of schizophrenia and in stress management, problem-solving, and social skills. Parents and siblings are included to gain knowledge and skills to support the adolescents.

The Self-Management Therapy intervention is administered in small multiple-family groups in 12 sessions over 7-1/2 months. The effects of the intervention on the patient and his/her family are assessed prior to treatment, after 6 sessions, after 12 sessions, and in a follow-up visit 6 months after completion of sessions.

A child may be eligible for this study if he/she:

Is 15 to 19 years old and has been diagnosed with schizophrenia.

DETAILED DESCRIPTION:
To test the effectiveness of a family-centered, community-based, self-management intervention (Self-Management Therapy) for adolescents with schizophrenia. The primary aim is to test its effectiveness in improving the adolescents' level of functioning in role performance, thinking/cognitive processing, behavior towards others, mood, and use of substances. The second aim is to assess the impact of the intervention on family functioning. The third aim is to describe the relationships among the process variables of the intervention.

Nakagawa-Kogan's self-management nursing model, Kanfer's self-regulation theory, and Liberman's theory of stress and vulnerability provide the theoretical basis for the self-management intervention developed specifically for a population with deficits in cognitive processing. The intervention involves training in symptom awareness, stress management skills, problem-solving, and social skills. Parents and siblings are included to gain knowledge and skills to support the adolescents.

The adolescent's level of functioning is assessed using the Child and Adolescent Functional Assessment Scale, the Birchwood Early Signs & Symptoms Scale for schizophrenia, and the DISA. Family Functioning is assessed by computing a Composite Family Functioning Index using weighted scores from the FACES II, Family Apgar, Family Empowerment, and Family Social Support scales. One parent is designated by the family to be the family respondent on the scales. The adolescents are referred to the study by mental health professionals. The intervention is administered in small multiple-family groups in 12 sessions over 7-1/2 months. Data are collected at 4 points in time: at baseline, after 6 intensive sessions, after 6 monthly reinforcement sessions, and 6 months post-intervention. ANCOVA is used to test the study hypotheses. Multivariate relationships are examined among the process variables of the intervention.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

Schizophrenia as diagnosed according to DSM-IV criteria when screened by a mental health professional using the K-SADS and the DISA.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 1998-04; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Increase in CAFAS level of functioning for all adolescents. | Over the course of 14 months

SECONDARY OUTCOMES:
Increase in family functioning for families in the treatment group according to the designated family respondent. | Over the course of 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen G. Schepp, PhD, Principal Investigator
Locations (1):
- University of Washington, Seattle, Washington, United States